CLINICAL TRIAL: NCT06100237
Title: Teclistamab or Talquetamab in Combination With Daratumumab SC for High-Risk Smoldering Myeloma: A Clinical and Correlative Phase 2 Sequential Cohort Immuno-Oncology Study to REVIVE Early Myeloma
Brief Title: Teclistamab or Talquetamab in Combination With Daratumumab for High-Risk Smoldering Myeloma (REVIVE Study)
Acronym: REVIVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carl Ola Landgren, MD, PhD (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Carl Ola Landgren, MD, PhD, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20221148
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Tec-Dara (Experimental): Participants will receive the recommended dosage combination treatment Tec-Dara.
  Interventions: Drug: Teclistamab; Drug: Daratumumab SC
- Cohort B: Tal-Dara (Experimental): Dosing and treatment schedule for participants in this group will be determined after Cohort A is completed.
  Interventions: Drug: Talquetamab; Drug: Daratumumab SC

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered by subcutaneous (SC) injection per discretion of treating physician. Participants will receive the recommended dosage.
  Arms: Cohort A: Tec-Dara
Drug: Talquetamab — Talquetamab will be administered per discretion of treating physician. Participants will receive the recommended dosage.
  Arms: Cohort B: Tal-Dara
Drug: Daratumumab SC — Daratumumab SC will be administered by subcutaneous (SC) injection per discretion of treating physician. Participants will receive the recommended dosage.

SUMMARY:
The purpose of this study is to see whether combination treatment of Teclistamab and Daratumumab (Tel-Dara) or combination Talquetamab and Daratumumab (Tal-Dara) will delay the onset of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed smoldering multiple myeloma (SMM) based on the IMWG Criteria10 including:

   * Serum M-protein ≥3 g/dL and/or BMPCs≥10 % (but <60%)
   * Absence of anemia: hemoglobin >10 g/dL
   * Absence of renal failure: serum creatinine <2.0 mg/dL
   * Absence of hypercalcemia: Calcium <10.5 mg/dL
   * Absence of lytic bone lesion on X-ray, CT, or positron emission tomography (PET)/CT and not more than 1 lesion on whole body MRI (NOTE: At the discretion of the Investigator, whole body CT or PET/CT may replace MRI in patients who have a contraindication or who are unable to have MRI performed.)
   * Involved/uninvolved light chain ratio <100 (unless involved light chain is ≤10 mg/dL) NOTE: Anemia, renal failure, and hypercalcemia is allowed if deemed unrelated to multiple myeloma (MM), see organ function criteria in point #5 below.
2. Patients must have measurable disease within the past 4 weeks, which is defined by any one of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL
   * Urine monoclonal protein >200 mg/24 hour
   * Serum immunoglobulin free light chain ≥10 mg/dL AND abnormal kappa/lambda serum free light chain ratio (reference: 0.26-1.65)
   * Other measurable disease as defined by the International Myeloma Working Group (IMWG).
   * Because the primary endpoint is MRD negativity based on bone marrow analysis, a patient without measurable disease in blood or urine may be enrolled and assessed for MRD negativity. NOTE: In patients who received minimal prior therapy within the allowable range per exclusion criteria 1, patients should have had documented measurable disease within 4 weeks of starting that respective therapy if currently unmeasurable.
3. Patients age ≥18 years.
4. Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0-1 assessed within the past 45 days. (See Appendix 17.1).
5. Patients must have adequate organ and marrow function ≤45 days as defined below:

   * Absolute neutrophil count (ANC) >1.0 K cells/μL; At the discretion of the Investigator, patients with an ANC of 0.5 K/μL-1.0 K/μL may also be enrolled if clinically appropriate (eg, patients with a baseline neutropenia that is chronic and/or ethnic neutropenia and that does not cause complications, e.g, no history of chronic infections).
   * Platelet count >75 K cells/μL
   * Hemoglobin >8 g/dL (transfusions are permissible if the cause of the anemia is other than myeloma)
   * Total bilirubin <1.5 X upper limit of normal (ULN). NOTE: Isolated total bilirubin ≥1.5 X ULN with conjugated [direct] bilirubin <1.5 X ULN is allowed for those participants with known Gilbert's syndrome.
   * Aspartate aminotransferase (AST)/ alanine transaminase (ALT) ≤2.5 X ULN
   * ≥30 mL/min based on Modification of Diet in Renal Disease (MDRD) 4-variable Formula calculation (Appendix 17.2) or creatine clearance (CrCl) measured by a 24-hour urine collection. The estimated glomerular filtration rate (eGFR) may also be determined by using other widely accepted methods as clinically indicated, ie, Cockcroft-Gault method or the chronic kidney disease (CKD)-epidemiology collaboration (EPI) per institutional standards.
6. Patients must have SMM that is categorized as high-risk for progression to MM-related end- organ damage by both clinical and genomic characteristics. Patients may be categorized as high risk by the Program for Study and Treatment of Malignant Hemopathies (PETHEMA) (immunoparesis and ≥95% aberrant bone marrow plasma cells (aBMPCs) by flow) and/or Mayo Clinic78 (20/2/20) criteria and/or have clonal BMPCs ≥10% with any one or more of the following criteria4:

   * Serum M protein ≥3 g/dL
   * Immunoglobulin A (IgA) SMM
   * Immunoparesis with reduction of 2 uninvolved immunoglobulin isotypes
   * Serum involved/uninvolved free light chain (FLC) ratio ≥8 (but <100)
   * Progressive increase in M-protein level (evolving type of SMM; increase in serum M- protein by ≥25% on 2 successive evaluations within a 6-month period)
   * Clonal bone marrow plasma cells (BMPC) 50%-59%
   * Abnormal plasma cell (PC) immunophenotype (≥95% of BMPCs are clonal) and reduction of ≥1 uninvolved immunoglobulin isotype(s)
   * Chromosomal abnormalities specifically translocation of chromosomes 4 or 14 (t(4;14)) or deletion of the short arm of chromosome 17 del(17p)) or gain of the long arm of chromosome 1 (1q gain) found in ≥5% of cells
   * Increased circulating PCs (PCs >5 x 106/L and/or >5% PCs per 100 peripheral blood mononuclear cells (PBMCs)
   * MRI with diffuse abnormalities or 1 focal lesion, AND/OR PET-CT with focal lesion with increased uptake without underlying osteolytic bone destruction.
7. A female participant of childbearing potential must have a negative serum or urine pregnancy test at screening (at or within 45 days of study enrollment) and within 72 hours of the start of study treatment (Section 4.7) and must agree to further serum or urine pregnancy tests during the study
8. A female participant must be (as defined in Appendix 17.3):

   1. Not of childbearing potential, or
   2. Of childbearing potential and practicing at least 1 highly effective method of contraception (see Appendix 17.3). NOTE: Participant must agree to continue the above throughout the study and for 3 months after the last dose of study treatment.

   NOTE: If a woman becomes of childbearing potential after start of the study, the woman must comply with point (b) as described above.
9. A female participant must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 3 months after receiving the last dose of study treatment. Female participants should consider preservation of eggs prior to study treatment, as anti-cancer treatments may impair fertility.
10. A female participant must agree to not breastfeed during the study and for a period of 5 months after receiving the last dose of study treatment.
11. A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for a period of 3 months after receiving the last dose of study treatment. If the male participant's partner is a female of childbearing potential, the male participant must use condoms (with or without spermicide), and the female partner of the male participant must also be practicing a highly effective method of contraception (see Appendix 17.3).

    NOTE: If the male participant is vasectomized, he still must wear a condom (with or without spermicidal foam/gel/film/cream/suppository), but his female partner is not required to use contraception.
12. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for period of 3 months after receiving the last dose of study treatment. Male participants should consider preservation of sperm prior to study treatment, as anti-cancer treatments may impair fertility.
13. Ability of the patient to understand and the willingness to sign a written informed consent document.
14. Have any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.
15. Must be willing and able to adhere to the lifestyle restrictions specified in this protocol (Section 3.3).

Exclusion Criteria:

1. Patients who have received prior systemic therapies for SMM/MM. One prior cycle (4-5 weeks) of therapy for SMM is allowed provided that patient undergoes a 4-week washout period prior to first dose of study treatment. Treatment with corticosteroids for other indications is permitted.
2. Patients who are receiving any other investigational agents for any reasons.
3. Patients who receive a live attenuated vaccine within 4 weeks of scheduled study treatment administration.
4. Contraindication to any concomitant medication, including those medications administered for infusion reaction, antiviral, antibacterial, anticoagulation, tumor lysis, or hydration prophylaxis given prior to therapy.
5. Patient has any of the following:

   1. Human immunodeficiency virus (HIV)-positive with 1 or more of the following:

      * History of acquired immune deficiency syndrome (AIDS)-defining conditions cluster of differentiation (CD4)count <350 cells/mm3
      * Detectable viral load during screening or within 6 months prior to screening
      * Not receiving highly active anti-retroviral therapy
      * Had a change in antiretroviral therapy within 6 months of the start of screening
      * Receiving antiretroviral therapy that may interfere with study treatment as assessed after discussion with the Medical Monitor
   2. Hepatitis B infection (ie, hepatitis B surface antigen (HBsAg) or hepatitis B virus (HBV)- DNA positive). Patients with resolved infection (ie, patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen (anti-HBc) and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV DNA levels. Those who are PCR positive will be excluded. In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status; see Section 10.3.5.2.1 for further required assessments.

      EXCEPTION: Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.
   3. Active hepatitis C infection as measured by positive HCV-ribonucleic acid (RNA) testing.

      Participants with a history of hepatitis C virus (HCV) antibody positivity must undergo HCV-RNA testing (Section 10.3.5.2.2). If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV-RNA positive) completed antiviral therapy and has undetectable HCV-RNA 12 weeks following the completion of therapy, the participant is eligible for the study.
   4. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for participants with known or suspected of having COPD or asthma, and participants must be excluded if FEV1 <50% of predicted normal.
   5. Moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification. Note that FEV1 testing is required for participants with known or suspected asthma, and participants must be excluded if FEV1 <50% of predicted normal.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the experimental agents used in study.
7. Female patient refuses to discontinue breastfeeding her infant during study treatment or within 5 months after receiving the last dose of study treatment.
8. Participant plans to father a child while enrolled in this study or within 3 months after the last dose of study treatment.
9. Presence of the following cardiac conditions:

   1. New York Heart Association stage III or IV congestive heart failure
   2. Myocardial infarction or coronary artery bypass graft ≤6 months prior to study enrollment
   3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
   4. Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities
   5. Unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina)
10. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, venous thromboembolic disease, hemorrhage, pulmonary fibrosis, pneumonitis, active autoimmune disease or a documented history of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing, or psychiatric illness/social situations within 2 weeks that would limit compliance with study requirements.
11. Active malignancy other than SMM requiring treatment in the past 24 months. Malignancies treated within the past 24 months that are considered cured with minimal risk of recurrence are allowed.
12. Have any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.
13. Patients with impaired decision-making capacity will not be enrolled on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) Negative as Measured by Flow Cytometry | 12 months
  MRD negative (10^-5 sensitivity by flow cytometry) as best response by completion of 12 cycles. MRD negative result means no disease is detected after treatment. Status of MRD will be assessed using International Myeloma Working Group (IMWG) Consensus Criteria for Response and Minimal Residual Disease Assessment in Multiple Myeloma, per discretion of treating physician.

SECONDARY OUTCOMES:
Number of Treatment Related Adverse Events | Up to 25 months
  The number of treatment related serious adverse events (SAEs) and grade 3 or higher adverse events (AEs) in participants receiving protocol therapy will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5, per physician discretion.
Overall Response Rate (ORR) | Up to 24 months
  Overall response rate (ORR) is determined by the number of participants achieving stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) to protocol therapy. Response will be assessed using standard International Myeloma Working Group (IMWG) Criteria for Response in Multiple Myeloma, per physician discretion.
Duration of Response (DoR) | Up to 24 months
  The duration of response (DoR) is measured as the time from when participants meet the criteria for stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) to protocol therapy using International Myeloma Working Group (IMWG) Criteria until the time progressive disease (PD) is documented, per discretion of treating physician.
Best Objective Responses (BoR) | Up to 24 months
  The rate of best objective responses (BoR) is determined by the number of participants who achieve stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) as their best response to protocol therapy using International Myeloma Working Group (IMWG) Criteria, per discretion of treating physician.
Minimal Residual Disease (MRD) Negativity Rate by Next-Generation Sequencing (NGS) | Up to 24 months
  The rate of minimal residual disease (MRD) negativity by next-generation sequencing (NGS) after 24 cycles of the protocol therapy is determined by the number of participants who achieve MRD negativity by 10^-6 sensitivity NGS, per discretion of treating physician.
Sustained MRD Negativity | Up to 7 years
  Sustained MRD negativity is determined by the number of participants who achieve MRD negativity 1, 2, and, 4 years apart, without any positive MRD in between, per discretion of treating physician.
Duration of MRD Negativity | Up to 7 years
  The duration of MRD negativity is measured as the time from the first time participants achieve MRD negativity until the participant has relapsed from MRD negativity, per discretion of treating physician.
Clinical progression-free survival (clinPFS) | Up to 7 years
  Clinical progression-free survival (clinPFS) is measured as the time from the participants start of protocol therapy to the clinical development of symptomatic multiple myeloma or death, per discretion of treating physician.
Biochemical progression-free survival (bioPFS) | Up to 7 years
  Biochemical progression-free survival (bioPFS) is measured as the time from the participants start of protocol therapy to progression of multiple myeloma in the blood or death occurs, using International Myeloma Working Group (IMWG) Criteria, per discretion of treating physician.
Overall Survival (OS) | Up to 7 years
  Overall Survival (OS) is determined by the amount of time from participants start of protocol therapy to death or to last known timepoint the participant was alive.
Serum Concentrations of Teclistamab and Talquetamab | Up to 7 years
  Serum samples will be analyzed to determine concentrations of Teclistamab and Talquetamab using validated, specific, and sensitive methods.
Pharmacokinetics of Teclistamab in multiple myeloma (MM) | Up to 7 years
  Serum from venous blood samples will be collected for measurement of serum concentrations of Teclistamab (Cohort A - Teclistamab only) and the generation of Anti-drug Antibodies (ADAs) where applicable to Teclistamab per the Study Schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Carl O Landgren, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No